CLINICAL TRIAL: NCT02107755
Title: A Phase 2 Study Using Stereotactic Ablative Radiation Therapy and Ipilimumab in Patients With Oligometastatic Melanoma
Brief Title: Stereotactic Radiation Therapy and Ipilimumab in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-12182; NCI-2014-00381 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Liver Metastases; Lung Metastases; Recurrent Melanoma; Stage IV Melanoma; Tumors Metastatic to Brain
Keywords: oligometastatic melanoma; melanoma
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (ipilimumab, stereotactic radiosurgery) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1 in weeks 1, 4, 7, and 10. Treatment repeats every 3 weeks for up to 4 total doses in the absence of disease progression or unacceptable toxicity. At approximately 5-6 weeks, patients undergo stereotactic radiosurgery over 2-3 days per week. Patients with stable disease or confirmed partial or complete response after completion of ipilimumab therapy at week 12 may receive re-induction ipilimumab at the discretion of the treating physician.
  Interventions: Biological: ipilimumab; Radiation: stereotactic radiosurgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Radiation: stereotactic radiosurgery — Undergo stereotactic radiosurgery
Other: laboratory biomarker analysis — Blood and tissue samples will be collected for research purposes.

SUMMARY:
This phase II trial studies the effectiveness of the combination of stereotactic radiation therapy and ipilimumab in patients with metastatic melanoma that has spread to four or fewer sites in the body (oligometastatic). Stereotactic radiation therapy is a type of external beam radiation therapy that uses special equipment to position the patient and precisely give a either a single large dose of radiation therapy to a tumor or several large doses of radiation therapy to a tumor using precision and accuracy that is guided by onboard daily imaging prior to radiation therapy. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some monoclonal antibodies find tumor cells and help kill them or carry tumor-killing substances to them. Giving stereotactic radiosurgery together with ipilimumab may kill more tumor cells by causing addition melanoma antigens to be presented to the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival of patients with oligometastatic melanoma treated with the combination of stereotactic ablative radiation therapy (SABR) (stereotactic radiosurgery) and ipilimumab in patients with oligometastatic melanoma using modified World Health Organization (mWHO) criteria.

SECONDARY OBJECTIVES:

I. To evaluate the 6-month progression-free survival of the combination of SABR and 3 mg/kg ipilimumab in patients with oligometastatic melanoma using immune related response criteria (irRC) criteria.

II. To evaluate the tolerability and safety of the combination. III. To evaluate the response rate based on mWHO & irRC criteria. IV. To evaluate the local control rate. V. To evaluate the overall survival rate.

TERTIARY OBJECTIVES:

I. Evaluate changes in blood and serum markers: absolute lymphocyte count, T-cell activation markers, T-cell suppression markers, T-helper cells and related cytokines, T-regulatory (T-reg) markers, co-stimulatory molecules, and serum cytokines when SABR is added to the ipilimumab regimen.

II. Evaluate genomic deoxyribonucleic acid (DNA) mutations in key melanoma genes and their correlation with response, progression-free survival, and overall survival.

OUTLINE:

Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1 in weeks 1, 4, 7, and 10. Treatment repeats every 3 weeks for up to 4 total doses in the absence of disease progression or unacceptable toxicity. At approximately 5-6 weeks, patients undergo stereotactic radiosurgery over 2-3 days per week. Patients with stable disease or confirmed partial or complete response after completion of ipilimumab therapy at week 12 may receive re-induction ipilimumab at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 30 and 90 days, every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histologic diagnosis of melanoma with metastatic disease to a visceral organ (lung, liver, brain, adrenal, nodal station outside the regional lymph drainage of the primary, vertebral bodies)
* 1-3 sites of metastatic disease able to be targeted by SABR
* White blood cells (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 75 x 10^3/uL
* Hemoglobin >= 9 g/dL (>= 80 g/L; may be transfused)
* Creatinine =< 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN for patients without liver metastasis, =< 5 times for liver metastases
* Bilirubin =< 2.0 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized

  * WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal; post-menopause is defined as:

    * Amenorrhea >= 12 consecutive months without another cause, or
    * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential
  * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab
  * Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Any other malignancy from which the patient has been disease-free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and Myasthenia Gravis)
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with ipilimumab or prior cluster of differentiation (CD)137 agonist or cytotoxic T-lymphocyte antigen 4 (CTLA-4) inhibitor or agonist
* A history of prior treatment with anti-programmed death (PD)-1 or anti-PD-L1 antibodies
* Concomitant therapy with any of the following: interleukin (IL)-2, interferon, other non-study immunotherapy regimens, cytotoxic chemotherapy, other investigation therapies
* Concomitant therapy with immune-suppressants or chronic use of systemic corticosteroids
* Must be off prior systemic therapies for 2 weeks prior to enrollment; patients that have been previously treated with systemic therapy adjuvantly or for metastatic disease remain eligible as long as they continue to meet all other eligibility criteria (oligometastatic, no visceral metastasis > 5 cm, eligible for SABR)
* Prior radiation therapy that at the treating physician's discretion makes SABR unsafe
* No evidence of pleural effusion or ascites
* Congestive heart failure > class II New York Heart Association (NYHA) or unstable angina
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Major surgery, open biopsy or significant traumatic injury within 2 weeks of first dose of study drug
* A visceral metastasis greater than 5 cm
* A visceral metastasis that due to its location cannot be safely treated with SABR
* Women of childbearing potential (WOCBP), defined above who:

  * Are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO)
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped
* Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized; before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy; all WOCBP MUST have a negative pregnancy test before first receiving ipilimumab; if the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bazan, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression-free Survival by mWHO Criteria
Description: Calculated along with corresponding 95% binomial confidence intervals. Kaplan-Meier curves will be used.
Time Frame: Time of study enrollment until the first documented date of disease progression, assessed up to 6 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 8
months | 0.75 [0.31 to 0.93]

2. Secondary Outcome: Rate of Progression-free Survival by irRC Criteria
Description: Calculated along with corresponding 95% binomial confidence intervals. Kaplan-Meier curves will be used.
Time Frame: Time of study enrollment until the first documented date of disease progression, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 8
months | 0.75 [0.31 to 0.93]

3. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Toxicities According to Common Toxicity Criteria for Adverse Events (CTCAE) Version 4
Description: Frequency and severity of adverse events and tolerability of the regimen in each of the patient groups will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: Up to 90 days after the last ipilimumab infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 8
Participants
  Alanine aminotransferase increased | 1
  Anemia | 1
  Aspartate aminotransferase increased | 1
  Diarrhea | 1
  Generalized muscle weakness | 1
  Hypernatremia | 1
  Hypertension | 1
  Lymphedema | 1
  Musculoskeletal and connective tissue disorder - Other, specify | 1
  Platelet count decreased | 1
  Rash maculo-papular | 1
  Thromboembolic event | 1
  Hyponatremia | 1

4. Secondary Outcome: Frequency of Objective Response Rate, Defined as Complete Response + Partial Response, Measured by Computed Tomography (CT) Using mWHO Criteria
Description: The response rate evaluated based on mWHO & irRC criteria
Time Frame: Up to 12 weeks
Population: Data was not collected and analyzed for the study
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of Objective Response Rate, Defined Using irRC
Time Frame: Up to 12 weeks
Population: Data was not collected and analyzed for the study
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Local Failure
Time Frame: Time of study enrollment until the first documented date of failure within the irradiated field, assessed up to 10 years
Population: Data was not collected and analyzed for the study
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Overall Survival
Description: Kaplan-Meier curves will be used.
Time Frame: Time of study enrollment until the time of death, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 8
months | 0.83 [0.27 to 0.97]

8. Other Pre Specified Outcome: Change in Marker Levels Between Those With vs. Without the Clinical Improvement
Description: Summarized univariately in a quantitative manner and also summarized by clinical outcome group (e.g. prog-free and alive at 6 months vs. not). Graphical analyses will be largely used to assess potential patterns and relationships; e.g. side-by-side boxplots to assess differences.
Time Frame: Baseline to week 50
Population: Data not collected and analyzed for the study
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of the study through the completion of the study which was up to an average of 5 years.
Description: The National Cancer Insitutes CTCAE version 4 was used to grade all adverse events.
Arm/Group | Treatment (Ipilimumab, Stereotactic Radiosurgery)
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab, Stereotactic Radiosurgery) (N=8)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Muscoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab, Stereotactic Radiosurgery) (N=8)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
Chills (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lymphedema (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02107755/Prot_SAP_000.pdf